CLINICAL TRIAL: NCT03884504
Title: A Prospective, Multi-Center, Single Arm Clinical Study to Evaluate the MDT-1118 Ventricular Assist Device System for Destination Therapy of Advanced Heart Failure
Brief Title: MDT-1118 Japan DT Study
Acronym: MDT-1118 Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT18052
Record Dates: First submitted 2019-03-15; First posted 2019-03-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure
Keywords: Advanced Heart Failure; Ventricular Assist Device System; Destination Therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ventricular Assist Device System — Ventricular Assist Device System

SUMMARY:
To evaluate the safety and effectiveness of the MDT-1118 VAD in a patient population for destination therapy (long term support) of advanced heart failure. The collected data will be used to support Japan regulatory application in expanding market approval for destination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥20 years of age at consent
2. In judgment of body size, body surface area (BSA) and anatomy by Investigator, patient can be implanted MDT-1118 VAD.
3. Patients with advanced heart failure symptoms (Class IIIB or IV) who are: (patient must meet one of the following)

   1. On optimal medical management, including dietary salt restriction and diuretics, for at least 45 out of the last 60 days and are failing to respond; or
   2. In Class III or Class IV heart failure for at least 14 days, and dependent on intra-aortic balloon pump (IABP) for 7 days and/or inotropes for at least 14 days
4. Left ventricular ejection fraction ≤ 25%
5. LVAD implant is intended as destination therapy
6. Must be able to receive the MDT-1118 VAD
7. Female patients of childbearing potential must agree to use adequate contraceptive precautions (defined as oral contraceptives, intrauterine devices, surgical contraceptives or a combination of condom and spermicide) for the duration of the study
8. The patient has signed the informed consent form and advance directive
9. The patient and the family understand that destination therapy is end-of-life medical care.

Exclusion Criteria:

1. Patients with INTERMACS profile 1
2. Existence of any ongoing mechanical circulatory support (MCS) other than an intra-aortic balloon pump (IABP)
3. Prior cardiac transplant
4. History of confirmed, untreated abdominal/ thoracic aortic aneurysm > 5 cm, or cardiac aneurysm or intraventricular septum rupture
5. Severe calcification in thoracic aorta
6. Cardiothoracic surgery within 14 days of implantation
7. Acute myocardial infarction within 14 days of implant as diagnosed by ST or T wave changes on the ECG, diagnostic biomarkers, ongoing pain and hemodynamic abnormalities as described in the guidelines published in ACC/AHA 2007 Guidelines for the Management of Patients with Unstable Angina/Non-ST-Elevation Myocardial Infarction1
8. Patients eligible for cardiac transplantation
9. On ventilator support for > 72 hours within the four days immediately prior to implantation
10. Pulmonary embolus within 21 days of implantation as documented by computed tomography (CT) scan or magnetic resonance imaging (MRI)
11. Symptomatic cerebrovascular disease, stroke within 180 days of implantation or > 80% stenosis of carotid or cranial vessels
12. Patient seems difficult to control device by oneself due to cerebral disorder
13. History of drug intoxication or alcohol dependence
14. Uncorrected moderate to severe aortic insufficiency. Correction may include repair or bioprosthesis at the time of implant
15. Severe right ventricular failure as defined by the anticipated need for right ventricular assist device (RVAD) support or extracorporeal membrane oxygenation (ECMO) at the time of screening or right atrial pressure > 20 mmHg on multiple inotropes or right ventricular ejection fraction (RVEF) <15% with clinical signs of severe right heart failure (e.g. Lower extremity edema, ascites or pleural effusions refractory to treatment with diuretics and two inotropic drugs)
16. Active, uncontrolled infection diagnosed by a combination of clinical symptoms and laboratory testing, including but not limited to, continued positive cultures, elevated temperature and white blood cell (WBC) count, hypotension, tachycardia, generalized malaise despite appropriate antibiotic, antiviral or antifungal treatment
17. Uncorrected thrombocytopenia or generalized coagulopathy (e.g., platelet count < 75,000, INR > 2.0 or PTT > 2.5 times control in the absence of anticoagulation therapy)
18. Intolerance to anticoagulant or antiplatelet therapies or any other peri- or postoperative therapy that the investigator may administer based upon the patient's health status
19. Serum creatinine > 3.0 mg/dL within 72 hours of implantation or requiring dialysis or ultrafiltration
20. Specific liver enzymes [AST (SGOT) and ALT (SGPT] > 3 times upper limit of normal within 72 hours of implantation
21. A total bilirubin > 3 mg/dL within 72 hours of implantation, or biopsy proven liver cirrhosis or portal hypertension
22. Patients with a mechanical heart valve
23. Etiology of heart failure is due to, or associated with, uncorrected thyroid disease, obstructive cardiomyopathy, pericardial disease, amyloidosis, active myocarditis or restrictive cardiomyopathy
24. History of severe COPD or severe restrictive lung disease (e.g FEV1 <50%) or severe pulmonary hypertension
25. Participation in any other study involving investigational drugs or devices
26. Severe illness, other than heart disease, which would limit survival to < 3 years
27. Peripheral vascular disease with rest pain or ischemic ulcers of the extremities
28. Pregnancy
29. Patient unwilling or unable to comply with study requirements
30. Technical obstacles, which pose an inordinately high surgical risk, in the judgment of the investigator
31. Inadequate family/social support
32. Systemic disease including collagen disease, insulin dependent severe diabetes or irreversible multi-organ failure.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Success at 12 months with the following definitions of success and failure | Implant to 12 months
  Therapy will be considered a success if, at the end of 12 months in the study:
  1. The subject is alive; and
  2. The subject has not had a stroke of Modified Rankin Score ≥ 4; and
  3. The subject retains the originally implanted device, unless the device was removed due to heart recovery, or the patient is electively transplanted.
  Therapy will be considered a failure if, within the 12 months in the study:
  1. The subject dies; or
  2. The subject has a stroke of Modified Rankin Score ≥ 4; or
  3. The device malfunctions or fails, requiring exchange, explantation, or urgent transplantation.

SECONDARY OUTCOMES:
Incidence of all adverse events per INTERMACS definition | Implant to 12 months
Incidence of all device malfunctions per INTERMACS definition | Implant to 12 months
Health Status improvement, as measured by KCCQ | Implant to 12 months
Health Status improvement, as measured by EuroQol EQ-5D-5L | Implant to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tokyo, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided